CLINICAL TRIAL: NCT06407219
Title: Evaluating and Improving Robot Assisted Gait Training
Brief Title: Evaluating the Impacts of a Single Session of Robot Assisted Gait Training With a Trexo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Elizabeth Condliffe, PhD MD, Assistant Clinical Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: REB21-1312
Record Dates: First submitted 2022-04-14; First posted 2024-05-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Physical Disability; CP (Cerebral Palsy); Developmental Disability
Keywords: Robot Assisted Gait Training; Trexo; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: This study is a randomized cross-over design, where participants will complete a training session in both the endurance mode and the strength mode of the Trexo robotic gait trainer. The session completed first will be randomized.
Who Masked: Participant
Masking Description: Participants will not know which mode they are completing on which day. Caregivers may be told if they ask, and investigators and outcome investigators will know the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive "Endurance" (Active Comparator): Participants will complete a training session using the Trexo robotic gait trainer in the "endurance" mode with a fixed gait pattern regardless of the participant's activity.
  Interventions: Device: Robot Assisted Gait Training
- Voluntary activity "Strength" (Active Comparator): Participants will complete a training session using the Trexo robotic gait trainer in the "strength" mode where the gait pattern is impacted by the participant's activity
  Interventions: Device: Robot Assisted Gait Training

INTERVENTIONS:
Device: Robot Assisted Gait Training — The Trexo robotic gait trainer will be used to facilitate physical activity in people who cannot walk independently, either at all or without the use of assistive gait aids (ie. walkers or canes). Session length will be determined by the participant's perceived fatigue level (ie. the session will run until the participant feels they want to or need to stop), and will not exceed 1 hour of training time.

SUMMARY:
Early use of robotic gait trainers have shown many benefits, however why these benefits occur and how to maximize them is unknown. There are a few options for how a robotic gait trainer can be used, however, there is not much understanding of how these options impact rehabilitation and compensate for impairments. The investigators aim to evaluate the impacts of as single session of Trexo robotic gait training and the impact of different modes of the Trexo robotic gait trainer. The investigators will evaluate how the different settings impact things like physical activity, walking, brain activity, spasticity, and fatigue. Investigators will arrange for a familiarity and fitting session to start, so that study team members can fit the participant to the Trexo and so that participants can become familiar with the feeling of using the Trexo robotic gait trainer. After the initial fitting sessions, follow up sessions will be completed to evaluate different settings on the Trexo, for example in "endurance" mode (where the robot completes the movements for the participant) and in "strength" mode (where the robot requires some assistance from the participant). Investigators may also test different fitting settings, for example with and without the supportive seat in the Trexo. Only three visits are required (one fitting/familiarity session and two testing sessions), however participants and/or their families may choose to complete more testing sessions if they want to assess other aspects of the training. For example, if the first two testing sessions assessed physical activity, participants and their families may choose to return for further sessions to assess brain activity. The aim of the study is to determine how robot assisted gait training impacts rehabilitation and compensates for impairments, as well as to provide suggestions on how the robotic gait trainer might be improved or modified. This study is exploratory to find out more about how these robotic gait trainers, specifically the Trexo, impacts various aspects of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Able to fit into the Trexo robotic gait trainer (<150 lbs., <5'7").
* Has impaired ability to walk due to a neurological or muscular disorder.

Exclusion Criteria:

* >150 lbs.
* >5'6" tall
* Medical contraindication to weight bearing (ie. recent orthopedic surgery)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Response to Exercise | Through study completion, an average of 4 weeks.
  We will use the collected heart rate as well as an estimated maximum heart rate (208-0.7*age) to determine the heart rate reserve (estimated maximum heart rate minus measured resting heart rate). Once the heart rate reserve has been calculated, the measured heart rate throughout the session will be used to determine how much time the participant spent above 40% of their heart rate reserve.

SECONDARY OUTCOMES:
Duration of Exercise Session | Through study completion, an average of 4 weeks.
  Total time participant spends actively using the Trexo. This is measured directly using the Trexo Robotics application.
Total Number of Steps Taken | Through study completion, an average of 4 weeks.
  Total number of steps that the participant takes in the robotic gait trainer for the duration of the session. This is measured directly in the Trexo Robotics application.
Average Number of Steps per Minute | Through study completion, an average of 4 weeks.
  Average number of steps taken per minute while actively using the Trexo. This is measured directly in the Trexo Robotics application.
Participant or Proxy Report of Rating of Perceived Exertion (RPE) | Through study completion, an average of 4 weeks.
  The participant's (or proxy, if participant is unable to communicate their RPE) perceived level of exertion for the robot assisted gait training session. This will be assessed using a rating of fatigue scale (0-10).
Brain Region Activation | Through study completion, an average of 4 weeks.
  Brain region activation will be assessed using electroencephalography (EEG) or functional near infrared spectroscopy (fNIRS). Both methods require participants to wear a cap in order to record this data. There are no contraindications to EEG or fNIRS.
Muscle Activation | Through study completion, an average of 4 weeks.
  Muscle activation will be assessed using electromyography (EMG) or mechanomyography (MMG). Both methods require surface electrodes to be placed on the skin. There are no contraindications to EMG or MMG.
Characteristics of Gait / Walking Pattern | Through study completion, an average of 4 weeks.
  Assessed using inertial measurement units (IMUs) during training sessions as well as between sessions to gather data on gait patterns outside of the robotic gait trainer. IMUs will be placed on the top of each foot of the participant (2 IMUs total).
Leg Muscle Spasticity | Through study completion, an average of 4 weeks.
  Assessed using the EMG/MMG (mentioned above) and the Biodex dynamometer. Muscles to be assessed may include: quadriceps, hamstrings, and plantarflexors. The leg will be moved passively through its range of motion while muscle activation is sensed using the sensors of the EMG/MMG system.
Physical Activity Level | Through study completion, an average of 4 weeks.
  Reported physical activity levels will be assessed using the habitual activity estimation scale (HAES) for a typical weekday as well as a typical weekend day. The HAES is a participant or proxy report of physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Condliffe, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada